CLINICAL TRIAL: NCT06566066
Title: Deep Geno- and Phenotyping of Patients With Thyroid Hormone Resistance, a Register Study.
Brief Title: Register for Patients With Thyroid Hormone Resistance.
Acronym: DEEPTYPE
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Markus Schuelke, M.D., Prof. Dr. med. Markus Schülke-Gerstenfeld, Charite University, Berlin, Germany
Other Study IDs: EA2_026_20
Record Dates: First submitted 2024-08-11; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Hypothyroidism; Global Developmental Delay; Intellectual Disability; Dystonia; Muscle Hypotonia; Seizures; Allan-Herndon-Dudley Syndrome; Microcephalus
Keywords: Thyroid hormone; Thyroid hormone resistance; MCT8; SLC16A2; THRA deficiency; Myelination
MeSH Terms: conditions — Hypothyroidism; Learning Disabilities; Intellectual Disability; Dystonia; Muscle Hypotonia; Seizures; Allan-Herndon-Dudley syndrome; Microcephaly; Thyroid Hormone Resistance Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with mutations in SLC16A2: Text
  Interventions: Other: no intervention
- Patients with mutations in THRA: Text
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — register study without intervention
  Other Names: does not apply

SUMMARY:
Thyroid hormones (TH) play a pivotal role in the development and function of the mammalian brain. Patients with impaired thyroid hormone transport into the brain tissue or in the case of defective local thyroid hormone receptor (collectively referred to as thyroid hormone resistance) subsequently experience psychomotor disabilities.

The "DEEPTYPE" registry has been established with the objective of intensifying the genotyping and, in particular, the neurological phenotyping of patients exhibiting deficiencies in either the thyroid hormone transporter (MCT8) or the thyroid hormone receptor alpha (THRα). The objective of this registry-based study is to enhance the diagnostic yield for MCT8 and THRα deficiencies by employing the serum fT3/fT4 ratio as a more sophisticated screening parameter. Furthermore, the investigators will study the genomic regulation of both genes and attempt to identify further coding and non-coding mutations that result in TH resistance. The patient registry "DEEPTYPE" will document the retrospective and prospective clinical data of identified children in a comprehensive manner. This will enable the identification of three key groups: (i) patients with non-coding mutations, (ii) patients with milder phenotypes presenting only with a subset of symptoms seen in both "classic" conditions, and (iii) patients who are ready for clinical trials.

DETAILED DESCRIPTION:
Thyroid hormones (TH) are of vital importance in the development and functioning of the brain. A deficiency in fetal thyroid hormone (TH) supply has been linked to significant psychomotor retardation in children born in regions with inadequate iodine supply. Insufficient postnatal production of thyroid hormones (TH) can result in intellectual and motor disabilities. These can be prevented by L-thyroxine (T4) supplementation in children with congenital hypothyroidism immediately after birth.

However, in the event of impaired transport of thyroid hormones into the brain tissue or in the case of defective local thyroid hormone receptors, the cerebral action of these hormones is impeded despite the presence of a sufficient thyroid hormone production. Such conditions may result from mutations in either SLC16A2, which encodes the monocarboxylate transporter 8 (MCT8), or THRA, which codes for the thyroid hormone receptor alpha (THRα). THRα is widely expressed in the central nervous system (CNS). In both instances, the absence of local TH action results in severe intellectual disability, developmental delay, movement disorders, and decreased brain volumes. In contrast to the outcomes observed in cases of congenital hypothyroidism, treatment trials involving the substitution of TH were ineffective in preventing the neurological phenotype in these children.

The full genotypic and phenotypic spectrum of these children has yet to be explored. It is anticipated that both conditions will be significantly underdiagnosed, given that awareness of these differential diagnoses within the pediatric community remains limited. As the standard screening parameters, such as thyroid-stimulating hormone (TSH), are not altered, the condition is frequently overlooked and is most often only "accidentally" diagnosed through next-generation sequencing.

The sole endocrine irregularity is a relative elevation of 3,3',5-triiodothyronine (T3) in comparison to T4. However, this is not a parameter that is routinely measured. More often the concentrations of the free plasma concentrations of these hormones, e.g. fT3 and fT4, are measured.

To date, only patients with mutations in the coding regions of the respective loci have been described. It can be reasonably assumed that mutations in the non-coding regulatory regions will result in disruption of the tissue-specific TH action in the MCT8/THRα-deficient brain. Similarly, disruptions in gene expression resulting from mutant regulatory enhancer sequences have recently been identified in other endocrine disorders, including congenital diabetes and brain developmental disorders.

The objective of this study is to enhance the diagnostic yield for MCT8 and THRα deficiencies by employing the serum fT3/fT4 ratio as a potentially more sophisticated screening parameter. Furthermore, the investigators will study the genomic regulation of both genes. The patient registry "DEEPTYPE" will be used to comprehensively document retrospective and prospective clinical data of identified children with coding or non-coding mutations. This will enable the investigators to identify patients with non-coding mutations and discover patients with milder phenotypes presenting only with a subset of symptoms seen in both "classic" conditions.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a coding or non-coding mutation in SLC16A2
* Presence of a coding or non-coding mutation in THRA
* Abnormal fT3/fT4 ratio in the serum
* Written informed consent of the caregivers for participation in the register study

Exclusion Criteria:

* Withdrawal of consent
* Correction/change of the molecular diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patients with THRα deficiency => Patients in whom a coding or non-coding pathogenic mutation was found in the THRA-gene or its regulating genomic regions (e.g. enhancers, promoters)
  * Patients with MCT8 deficiency => Patients in whom a coding or non-coding pathogenic mutation was found in the SLC16A2-gene or its regulating genomic regions (e.g. enhancers, promoters)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2029-07-14 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Description of infant motor and language development | 5 years
  Bayley Scales of Infant and Toddler Development III => (Units on a Scale and Sum Score)
Description of neurological abnormalities | 5 years
  Hammersmith Infant Neurological Examination (HINE) => (Units on a Scale and Sum Score)
Description of motor development | 5 years
  Gross Motor Function Measure (GMFM-88) => (Units on a Scale and Sum Score)

SECONDARY OUTCOMES:
body weight | 5 years
  kilograms
body length | 5 years
  centimeters
head circumference | 5 years
  centimeters
Reponse to therapies (e.g. Triac, DIPTA, levodopa/carbidopa) | 5 years
  Recording of responses to standard and experimental therapies
T3 | 5 years
  microgram per liter
T4 | 5 years
  microgram per liter
fT3 | 5 years
  microgram per liter
fT4 | 5 years
  microgram per liter
TSH | 5 years
  mU per litre
CSF fT3 | 5 years
  microgram per liter
CSF fT4 | 5 years
  microgram per liter
CSF levodopa | 5 years
  micromol/l
CSF homovanillic acid (HVA) | 5 years
  micromol/l
CSF 5-hydroxyindoleacetic acid (5-HIAA) | 5 years
  micromol/l
Quantification of dystonia | 5 years
  Burke-Fahn-Marsden Dystonia Rating Scale => (Units on a Scale and Sum Score)
Quantification of parkinsonism in children | 5 years
  Parkinsonism Dystonia Scale for Infants and Young Children => (Units on a Scale and Sum Score)
Quanitification of cerebral palys symptomes | 5 years
  Cerebral Palsy Child Health Index of Life with Disabilities => (Units on a Scale and Sum Score)

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Krude, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charite - Universitaetsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wilpert NM, Krueger M, Opitz R, Sebinger D, Paisdzior S, Mages B, Schulz A, Spranger J, Wirth EK, Stachelscheid H, Mergenthaler P, Vajkoczy P, Krude H, Kuhnen P, Bechmann I, Biebermann H. Spatiotemporal Changes of Cerebral Monocarboxylate Transporter 8 Expression. Thyroid. 2020 Sep;30(9):1366-1383. doi: 10.1089/thy.2019.0544. Epub 2020 Apr 17. PMID 32143555
- [Background] Friesema EC, Grueters A, Biebermann H, Krude H, von Moers A, Reeser M, Barrett TG, Mancilla EE, Svensson J, Kester MH, Kuiper GG, Balkassmi S, Uitterlinden AG, Koehrle J, Rodien P, Halestrap AP, Visser TJ. Association between mutations in a thyroid hormone transporter and severe X-linked psychomotor retardation. Lancet. 2004 Oct 16-22;364(9443):1435-7. doi: 10.1016/S0140-6736(04)17226-7. PMID 15488219
- [Background] Remerand G, Boespflug-Tanguy O, Tonduti D, Touraine R, Rodriguez D, Curie A, Perreton N, Des Portes V, Sarret C; RMLX/AHDS Study Group. Expanding the phenotypic spectrum of Allan-Herndon-Dudley syndrome in patients with SLC16A2 mutations. Dev Med Child Neurol. 2019 Dec;61(12):1439-1447. doi: 10.1111/dmcn.14332. Epub 2019 Aug 13. PMID 31410843
- [Background] Groeneweg S, Peeters RP, Moran C, Stoupa A, Auriol F, Tonduti D, Dica A, Paone L, Rozenkova K, Malikova J, van der Walt A, de Coo IFM, McGowan A, Lyons G, Aarsen FK, Barca D, van Beynum IM, van der Knoop MM, Jansen J, Manshande M, Lunsing RJ, Nowak S, den Uil CA, Zillikens MC, Visser FE, Vrijmoeth P, de Wit MCY, Wolf NI, Zandstra A, Ambegaonkar G, Singh Y, de Rijke YB, Medici M, Bertini ES, Depoorter S, Lebl J, Cappa M, De Meirleir L, Krude H, Craiu D, Zibordi F, Oliver Petit I, Polak M, Chatterjee K, Visser TJ, Visser WE. Effectiveness and safety of the tri-iodothyronine analogue Triac in children and adults with MCT8 deficiency: an international, single-arm, open-label, phase 2 trial. Lancet Diabetes Endocrinol. 2019 Sep;7(9):695-706. doi: 10.1016/S2213-8587(19)30155-X. Epub 2019 Jul 31. PMID 31377265
- [Background] Groeneweg S, van Geest FS, Abaci A, Alcantud A, Ambegaonkar GP, Armour CM, Bakhtiani P, Barca D, Bertini ES, van Beynum IM, Brunetti-Pierri N, Bugiani M, Cappa M, Cappuccio G, Castellotti B, Castiglioni C, Chatterjee K, de Coo IFM, Coutant R, Craiu D, Crock P, DeGoede C, Demir K, Dica A, Dimitri P, Dolcetta-Capuzzo A, Dremmen MHG, Dubey R, Enderli A, Fairchild J, Gallichan J, George B, Gevers EF, Hackenberg A, Halasz Z, Heinrich B, Huynh T, Klosowska A, van der Knaap MS, van der Knoop MM, Konrad D, Koolen DA, Krude H, Lawson-Yuen A, Lebl J, Linder-Lucht M, Lorea CF, Lourenco CM, Lunsing RJ, Lyons G, Malikova J, Mancilla EE, McGowan A, Mericq V, Lora FM, Moran C, Muller KE, Oliver-Petit I, Paone L, Paul PG, Polak M, Porta F, Poswar FO, Reinauer C, Rozenkova K, Menevse TS, Simm P, Simon A, Singh Y, Spada M, van der Spek J, Stals MAM, Stoupa A, Subramanian GM, Tonduti D, Turan S, den Uil CA, Vanderniet J, van der Walt A, Wemeau JL, Wierzba J, de Wit MY, Wolf NI, Wurm M, Zibordi F, Zung A, Zwaveling-Soonawala N, Visser WE. Disease characteristics of MCT8 deficiency: an international, retrospective, multicentre cohort study. Lancet Diabetes Endocrinol. 2020 Jul;8(7):594-605. doi: 10.1016/S2213-8587(20)30153-4. PMID 32559475
- [Background] Tonduti D, Vanderver A, Berardinelli A, Schmidt JL, Collins CD, Novara F, Genni AD, Mita A, Triulzi F, Brunstrom-Hernandez JE, Zuffardi O, Balottin U, Orcesi S. MCT8 deficiency: extrapyramidal symptoms and delayed myelination as prominent features. J Child Neurol. 2013 Jun;28(6):795-800. doi: 10.1177/0883073812450944. Epub 2012 Jul 17. PMID 22805248
- [Result] Masnada S, Sarret C, Antonello CE, Fadilah A, Krude H, Mura E, Mordekar S, Nicita F, Olivotto S, Orcesi S, Porta F, Remerand G, Siri B, Wilpert NM, Amir-Yazdani P, Bertini E, Schuelke M, Bernard G, Boespflug-Tanguy O, Tonduti D. Movement disorders in MCT8 deficiency/Allan-Herndon-Dudley Syndrome. Mol Genet Metab. 2022 Jan;135(1):109-113. doi: 10.1016/j.ymgme.2021.12.003. Epub 2021 Dec 16. PMID 34969638
- [Result] Wilpert NM, Tonduti D, Vaia Y, Krude H, Sarret C, Schuelke M. Establishing Patient-Centered Outcomes for MCT8 Deficiency: Stakeholder Engagement and Systematic Literature Review. Neuropsychiatr Dis Treat. 2023 Oct 20;19:2195-2216. doi: 10.2147/NDT.S379703. eCollection 2023. PMID 37881807